CLINICAL TRIAL: NCT05451914
Title: My Diabetes Care: A Pragmatic, Parallel-design, Randomized Controlled Trial
Brief Title: Effects of My Diabetes Care on Patient Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, William Martinez, MD, MS, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 230106; R01DK131129 (NIH)
Record Dates: First submitted 2022-07-01; First posted 2022-07-11 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Patient Web Portals; Health Information Technology
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- My Diabetes Care (Experimental): Patients have access to an existing patient web portal (i.e., Epic's MyChart) embedded with My Diabetes Care.
  Interventions: Other: My Diabetes Care
- Usual Care (No Intervention): Patients will have access to an existing patient web portal (i.e., Epic's MyChart) NOT embedded with My Diabetes Care (i.e., usual care)

INTERVENTIONS:
Other: My Diabetes Care — My Diabetes Care (MDC) is a multi-faceted patient portal intervention for mobile devices that is designed to help patients better understand their diabetes health data as well as promote and support self-management. MDC uses infographics to facilitate patients' understanding of their diabetes health data (e.g., HbA1c, LDL) and provides literacy level-appropriate and tailored diabetes self-care information.
  Other Names: Patient-facing Diabetes Dashboard
  Arms: My Diabetes Care

SUMMARY:
The purpose of this study is to conduct a two-arm, parallel-design, pragmatic randomized controlled trial of a patient portal intervention for diabetes, My Diabetes Care (MDC), to evaluate its effect on clinical outcomes.

DETAILED DESCRIPTION:
484 adult patients with type 2 diabetes mellitus will be randomized to one of two arms. 242 will be assigned to the intervention (My Diabetes Care) embedded within an existing patient web portal, My Health at Vanderbilt at Vanderbilt University Medical Center or Patient Gateway at Brigham and Women's Hospital. 242 will be assigned to a usual care comparison arm with access currently available version of My Health at Vanderbilt or Patient Gateway without the My Diabetes Care (MDC) application. Potentially eligible patients will be invited to be screened for enrollment in the study. Interested patients will be able to complete an electronic consent form and enroll online via Research Electronic Data Capture (REDCap). Outcomes data will be collected from patients at four time points: baseline (T0), three-month follow-up (T1), three-month follow-up (T2), six-month follow-up (T3), and twelve-month follow-up (T4). At each time point, study participants will complete questionnaires electronically via email using REDCap, participants' hemoglobin A1C level will be assess via home A1C test kits, and participants' diabetes health data will be abstracted from their electronic health record. Participants will be randomized to the intervention or control arm after their baseline data is collected.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* Age 18-75 years old
* Currently taking at least one medication for diabetes
* Be a patient at Vanderbilt University Medical Center (VUMC) or Brigham and Women's Hospital (BWH)
* Able to speak and read in English or Spanish
* Have reliable access to a smartphone, tablet, or computer with internet access
* Active patient web portal account (My Health at Vanderbilt at VUMC or Patient Gateway at BWH)

Exclusion Criteria:

* Receiving dialysis,
* Pregnant or planning to become pregnant within the next year,
* Living in a long-term care facility.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Change in Blood Glucose Control | Baseline (T0), Three-month Follow-up (T1), Six-month Follow-Up (T2), Twelve-month Follow-up (T3)
  Hemoglobin A1c will assessed using mail-in home HbA1c test kits and participants' most recent hemoglobin A1C will be abstracted from participants' electronic medical record.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline (T0), Three-month Follow-up (T1), Six-month Follow-Up (T2), Twelve-month Follow-up (T3)
  Participants' most recent body mass index (BMI) measurement will be abstracted from participants' electronic medical record.
Change in Low Density Lipoprotein (LDL) | Baseline (T0), Three-month Follow-up (T1), Six-month Follow-Up (T2), Twelve-month Follow-up (T3)
  Participants' most recent low density lipoprotein (LDL) measurement will be abstracted from participants' electronic medical record.
Urine Albumin-to-Creatinine Ratio | Baseline (T0), Three-month Follow-up (T1), Six-month Follow-Up (T2), Twelve-month Follow-up (T3)
  Participants' most albumin-to-creatinine ratio will be abstracted from participants' electronic medical record.
Change in Blood Pressure Control | Baseline (T0), Three-month Follow-up (T1), Six-month Follow-Up (T2), Twelve-month Follow-up (T3)
  Participants' most recent blood pressure measurement will be abstracted from participants' electronic medical record and will be used to calculate the participants' mean arterial pressure (MAP) using the following formula: MAP = diastolic pressure + 1/3(systolic pressure - diastolic pressure).
Change in Diabetes Self-Care (General Diet Adherence) | Baseline (T0), Three-month Follow-up (T1), Six-month Follow-Up (T2), Twelve-month Follow-up (T3)
  The Summary of Diabetes Self-Care Activity (SDSCA) is a 10-item multidimensional instrument to assess levels of diabetes self-care across five domains: general diet (2 items), specific diet (2 items), exercise (2 items), foot care (2 items), and blood-glucose testing (2 items). The general diet subscale is used to assess general diet adherence. The instrument is based on the self-reported days completing recommended activities during the past 7 days. An example item includes "How many of the last SEVEN DAYS have you followed a healthful eating plan?" The general diet subscale score is the mean number of days for the 2 items in the subscale. The score range is from 0 days (worst) to 7 days (best).
Change in Diabetes Self-Care (Exercise Adherence) | Baseline (T0), Three-month Follow-up (T1), Six-month Follow-Up (T2), Twelve-month Follow-up (T3)
  The Summary of Diabetes Self-Care Activity (SDSCA) is a 10-item multidimensional instrument to assess levels of diabetes self-care across five domains: general diet (2 items), specific diet (2 items), exercise (2 items), foot care (2 items), and blood-glucose testing (2 items). The exercise subscale is used to assess exercise adherence. The instrument is based on the self-reported days completing recommended activities during the past 7 days. An example item includes "On how many of the last SEVEN DAYS did you participate in at least 30 minutes of physical activity?" The exercise subscale score is the mean number of days for the 2 items in the subscale. The score range is from 0 days (worst) to 7 days (best).
Change in Diabetes Self-Care (Diabetes Medication Adherence) | Baseline (T0), Three-month Follow-up (T1), Six-month Follow-Up (T2), Twelve-month Follow-up (T3)
  The Adherence to Refills and Medications Scale-Diabetes (ARMS-D) is a reliable and valid measure of diabetes medication adherence. The 11-item ARMS-D has good internal consistency reliability (α=0.86). Responses range from 1="none of the time" to 4="all of the time," and are summed to produce an overall adherence score ranging from 12-48, with higher scores representing more problems with medication adherence.
Change in Diabetes Self-Care (Self-Monitoring of Blood Glucose Adherence) | Baseline (T0), Three-month Follow-up (T1), Six-month Follow-Up (T2), Twelve-month Follow-up (T3)
  The Summary of Diabetes Self-Care Activity (SDSCA) is a 10-item multidimensional instrument to assess levels of diabetes self-care across five domains: general diet (2 items), specific diet (2 items), exercise (2 items), foot care (2 items), and blood-glucose testing (2 items). The blood-glucose testing subscale is used to assess self-monitoring of blood glucose adherence. The instrument is based on the self-reported days completing recommended activities during the past 7 days. An example item includes "On how many of the last SEVEN DAYS did you test your blood sugar?" The blood-glucose testing subscale is the mean number of days for the 2 items in the subscale. The score range is from 0 days (worst) to 7 days (best).
Usability of MyChart (for Control Group) | Baseline (T0), Three-month Follow-up (T1), Six-month Follow-Up (T2), Twelve-month Follow-up (T3)
  The usability of the patient portal (Epic's MyChart) will be assessed using the System Usability Scale (SUS). The SUS is a valid measure of usability and assesses users' perceptions of ease of use, likability of the interface, and overall satisfaction using a 5- point Likert scale (strongly disagree to strongly agree). The ten items are scored on a five-point Likert scale. The item scores are summed and then converted to a score ranging from 0 (worst) to 100 (best). Based on prior research, a score above 68 would be above average and a score of 85 or above suggests excellent usability.
Satisfaction/Usability of My Diabetes Care (for Intervention Group) | Baseline (T0), Three-month Follow-up (T1), Six-month Follow-Up (T2), Twelve-month Follow-up (T3)
  The usability of the My Diabetes Care will be assessed using the System Usability Scale (SUS). The SUS is a valid measure of usability and assesses users' perceptions of ease of use, likability of the interface, and overall satisfaction using a 5- point Likert scale (strongly disagree to strongly agree). The ten items are scored on a five-point Likert scale. The item scores are summed and then converted to a score ranging from 0 (worst) to 100 (best). Based on prior research, a score above 68 would be above average and a score of 85 or above suggests excellent usability.

CONTACTS AND LOCATIONS:
Overall Officials: William Martinez, MD, MS, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
After study results are posted on clinical trials and published in a peer-reviewed journal, de-identified individual participant data that underlie the results reported will be available upon requests made to the principal investigator and ending after 36 months after publication.
Supporting Information: Study Protocol, SAP
Time Frame: Deidentified individual participant data that underlie the results reported will be available after publication in a peer-reviewed journal and posted on clinical trials and ending after 36 months of publication.
Access Criteria: Researchers should provide a methodologically sound proposal to achieve their proposed aims. Proposals may be submitted to the principal investigator up to 36 months following publication. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2024-07-26): https://cdn.clinicaltrials.gov/large-docs/14/NCT05451914/ICF_000.pdf